CLINICAL TRIAL: NCT07407400
Title: Lemborexant for Sleep Promotion and Delirium Prevention in Critically Ill Adults: A Combined Feasibility-Pilot, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Lemborexant for Sleep and Delirium Prevention in Elderly ICU Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEM-SICU
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Sleep Disturbance; Delirium; Critical Illness
Keywords: Lemborexant; Dual Orexin Receptor Antagonist; Sleep Disturbance; Delirium; Intensive Care Unit; Critically Ill Elderly
MeSH Terms: conditions — Parasomnias; Delirium; Critical Illness | interventions — lemborexant

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to receive either lemborexant or matching placebo. Each participant receives only one assigned intervention and is followed in parallel for study outcomes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study medication (lemborexant and placebo) is over-encapsulated to appear identical. Participants, bedside clinical staff, investigators, outcome assessors, and data analysts are blinded to treatment allocation. Emergency unblinding is available through the hospital pharmacy if clinically required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lemborexant (Experimental): Participants receive lemborexant 2.5 mg (half of a 5-mg tablet) administered orally or via nasogastric tube once nightly at 20:00 ± 30 minutes for three consecutive nights. All participants also receive standard non-pharmacologic sleep-promoting care in the ICU.
  Interventions: Drug: Lemborexant
- Placebo (Placebo Comparator): Participants receive a matching placebo administered orally or via nasogastric tube once nightly at 20:00 ± 30 minutes for three consecutive nights. All participants also receive standard non-pharmacologic sleep-promoting care in the ICU.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lemborexant — Lemborexant is administered at a dose of 2.5 mg (half of a 5-mg tablet) once nightly at 20:00 ± 30 minutes for three consecutive nights. The medication is given orally or via nasogastric tube. For nasogastric administration, the tablet is crushed, mixed with sterile water, and flushed through the tube. Lemborexant is over-encapsulated to maintain blinding. All participants also receive standard non-pharmacologic sleep-promoting care in the ICU, including light reduction, noise and alarm adjustment, and clustering of care.
  Arms: Lemborexant
Drug: Placebo — A matching inert placebo tablet/capsule identical in appearance to lemborexant is administered orally or via nasogastric tube once nightly at 20:00 ± 30 minutes for three consecutive nights. The placebo is over-encapsulated to maintain blinding. All participants receive standard non-pharmacologic sleep-promoting care in the ICU, including light reduction, noise and alarm adjustment, and clustering of care.
  Arms: Placebo

SUMMARY:
Sleep disturbance is very common among critically ill patients in the intensive care unit (ICU), particularly in older adults after surgery. Poor sleep in the ICU is associated with important complications, including delirium, longer duration of mechanical ventilation, prolonged hospital stay, and increased mortality. Current non-drug approaches to improve sleep, such as reducing noise and light and clustering nursing care, may provide limited benefit and are often difficult to implement consistently. Safe and effective drug treatments for sleep in critically ill older patients remain limited.

Lemborexant is a dual orexin receptor antagonist that promotes sleep by blocking wake-promoting pathways in the brain. Unlike many traditional sleep medications, lemborexant has minimal effects on breathing and has been shown to be well tolerated in older adults with insomnia. However, its effects on sleep and delirium have not been studied in critically ill patients.

This study is a single-center, randomized, double-blind, placebo-controlled feasibility and pilot trial conducted in the surgical intensive care unit of Siriraj Hospital, Bangkok, Thailand. The study will enroll 100 critically ill postoperative patients aged 65 years or older who are expected to remain in the ICU for at least 48 hours. Participants will be randomly assigned to receive either low-dose lemborexant (2.5 mg) or a matching placebo once nightly for three consecutive nights. All participants will also receive standard non-pharmacologic sleep-promoting care used in the ICU.

The main goals of this pilot study are to evaluate the feasibility and safety of administering lemborexant in elderly ICU patients and to explore its potential effects on sleep and delirium. Sleep will be assessed using both subjective questionnaires completed each morning and objective wrist-worn actigraphy to measure sleep duration and sleep stages. Delirium will be assessed twice daily using a standardized delirium screening tool for up to seven days or until ICU discharge. Additional outcomes include medication adherence, adverse events, duration of mechanical ventilation, length of ICU and hospital stay, and in-hospital mortality.

The results of this study will provide important preliminary data on the feasibility, safety, and potential benefits of lemborexant in critically ill older adults and will help inform the design of future larger clinical trials aimed at improving sleep and reducing delirium in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older.
* Admission to the Surgical Intensive Care Unit (SICU).
* Anticipated ICU stay of at least 48 hours, as assessed by the ICU consultant and responsible surgeon.
* Able to receive enteral medication via oral or nasogastric route.

Exclusion Criteria:

* Requirement for frequent neurological checks or scheduled awakening (e.g., acute stroke or neurosurgery).
* Deep sedation defined as Richmond Agitation-Sedation Scale (RASS) ≤ -3.
* Positive Confusion Assessment Method for the ICU (CAM-ICU) within 12 hours prior to randomization.
* Severe hemodynamic or respiratory instability requiring neuromuscular blockers or high-dose vasopressors (e.g., norepinephrine ≥ 0.1 µg/kg/min and titrating upward).
* High risk of aspiration, including ongoing vomiting, gastric residual volume >250 mL, or intolerance to oral or enteral medications.
* Concomitant use of strong CYP3A inhibitors or inducers (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, rifampicin, carbamazepine, phenytoin, or St. John's wort).
* Severe hepatic impairment (Child-Pugh class C).
* End-stage kidney disease or chronic kidney disease stage 5.
* Concomitant use of sedative-hypnotic medications, including benzodiazepines, Z-drugs, trazodone, tricyclic antidepressants, melatonin, or other sleep-inducing agents.
* Known hypersensitivity to lemborexant or other dual orexin receptor antagonists.
* History of cataplexy-like symptoms or severe depression with suicidal ideation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time Assessed by Actigraphy | Nights 1-3 of the intervention period (20:00 to 08:00 each night)
  Total sleep time (TST) measured using wrist-worn actigraphy (Fitbit Charge 5), defined as the total number of minutes scored as sleep during the nighttime period.

SECONDARY OUTCOMES:
Subjective Sleep Quality Assessed by Richards-Campbell Sleep Questionnaire | Each morning after Nights 1-3 of the intervention period (approximately 08:00)
  Subjective Sleep Quality Assessed by the Richards-Campbell Sleep Questionnaire (RCSQ).
  Subjective sleep quality will be assessed using the validated Thai version of the Richards-Campbell Sleep Questionnaire. The RCSQ consists of five items (sleep depth, sleep latency, number of awakenings, efficiency of returning to sleep, and overall sleep quality), each rated on a visual analogue scale ranging from 0 to 50 mm, where 0 represents the poorest sleep and 50 represents the best sleep. The total RCSQ score is calculated as the mean of the five item scores, yielding a composite score ranging from 0 to 50, with higher scores indicating better subjective sleep quality.
Delirium Incidence Assessed by CAM-ICU | From randomization until ICU Day 7 or ICU discharge, whichever occurs first
  Delirium incidence will be assessed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), a validated diagnostic instrument for delirium in critically ill patients. The CAM-ICU is not a continuous or ordinal scale but a binary diagnostic assessment, yielding either a positive (delirium present) or negative (delirium absent) result based on four core features (acute change or fluctuating course, inattention, altered level of consciousness, and disorganized thinking).
  Delirium incidence is defined as the occurrence of at least one positive CAM-ICU assessment during the observation period. As this outcome is dichotomous, minimum and maximum scale values are not applicable, and higher or lower scores do not represent better or worse outcomes.
Delirium Duration | From randomization until ICU Day 7 or ICU discharge, whichever occurs first
  Delirium duration defined as the total number of days with a positive CAM-ICU assessment during the observation period.
Objective Sleep Stage Proportions Assessed by Actigraphy | Nights 1-3 of the intervention period (20:00 to 08:00 each night)
  Objective sleep architecture will be assessed using wrist-worn actigraphy (Fitbit Charge 5). Sleep stage proportions, including deep sleep, light sleep, and rapid eye movement (REM) sleep, will be derived from actigraphy algorithms and expressed as the percentage (%) of total sleep time for each night.
  Each sleep stage proportion ranges from 0% to 100%, where higher values indicate a greater proportion of time spent in that specific sleep stage. No composite or total score is calculated for this outcome.
Composite Sleep Score Assessed by Actigraphy | Nights 1-3 of the intervention period (20:00 to 08:00 each night).
  Overall objective sleep quality will be assessed using the composite sleep score generated by wrist-worn actigraphy (Fitbit Charge 5). The composite sleep score is a proprietary summary metric derived from multiple actigraphy-based parameters, including sleep duration, continuity, and sleep stage distribution.
  The composite sleep score ranges from 0 to 100, where higher scores indicate better overall objective sleep quality.
Safety and Adverse Events | From the first dose of study medication until ICU discharge, assessed for up to 7 days after randomization, whichever occurs first.
  Safety will be assessed by the frequency and nature of adverse events (AEs) and serious adverse events (SAEs) potentially related to the study medication. Prespecified events of interest include oversedation, respiratory compromise, aspiration, and excessive somnolence. Adverse events will be identified through daily clinical assessment and review of medical records and recorded according to standard ICU reporting practices.
  This outcome is descriptive and categorical. It is not based on a numerical scale, and minimum or maximum values are not applicable.
Recruitment Rate | During the recruitment period, from first patient screened to last patient randomized.
  Recruitment rate will be assessed as the proportion of eligible patients who are successfully enrolled and randomized into the study during the recruitment period. The recruitment rate is calculated as the number of randomized participants divided by the total number of eligible patients screened.
  The recruitment rate ranges from 0% to 100%, with higher values indicating greater feasibility of patient enrollment.
Medication Adherence to Study Drug | Nights 1-3 of the intervention period
  Medication adherence will be assessed as the proportion of prescribed study drug doses that are successfully administered during the intervention period. Adherence will be determined from medication administration records.
  Medication adherence is expressed as a percentage (%) of planned doses received, ranging from 0% to 100%, where higher values indicate better adherence.
Completion Rate of Subjective Sleep Assessments | Each morning after Nights 1-3 of the intervention period (approximately 08:00).
  Completion of subjective sleep assessments will be assessed as the proportion of expected Richards-Campbell Sleep Questionnaire (RCSQ) assessments that are completed by participants.
  The completion rate ranges from 0% to 100%, with higher values indicating better feasibility of questionnaire-based sleep assessment.
Adequacy of Actigraphy Wear Time | Nights 1-3 of the intervention period (20:00 to 08:00 each night).
  Adequacy of actigraphy wear time will be assessed using wrist-worn actigraphy (Fitbit Charge 5) and defined as the proportion of nights with valid actigraphy data, according to prespecified criteria for minimum wear duration during the sleep period.
  Adequacy is expressed as a percentage (%) of monitored nights with valid data, ranging from 0% to 100%, where higher values indicate better feasibility of actigraphy-based sleep monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Nuanprae Kitisin, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Mahidol University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitisin N, Somnuke P, Thikom N, Raykateeraroj N, Poontong N, Thanakiattiwibun C, Wongtangman K. Psychometric properties of a Thai version of the Richards-Campbell sleep questionnaire. Nurs Crit Care. 2022 Nov;27(6):885-892. doi: 10.1111/nicc.12705. Epub 2021 Aug 23. PMID 34425024
- [Background] Tilouche N, Hassen MF, Ali HBS, Jaoued O, Gharbi R, El Atrous SS. Delirium in the Intensive Care Unit: Incidence, Risk Factors, and Impact on Outcome. Indian J Crit Care Med. 2018 Mar;22(3):144-149. doi: 10.4103/ijccm.IJCCM_244_17. PMID 29657370
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Drouot X, Cabello B, d'Ortho MP, Brochard L. Sleep in the intensive care unit. Sleep Med Rev. 2008 Oct;12(5):391-403. doi: 10.1016/j.smrv.2007.11.004. Epub 2008 May 23. PMID 18502155
- [Background] Parthasarathy S, Tobin MJ. Sleep in the intensive care unit. Intensive Care Med. 2004 Feb;30(2):197-206. doi: 10.1007/s00134-003-2030-6. Epub 2003 Oct 16. PMID 14564378